CLINICAL TRIAL: NCT01836328
Title: Prospective Randomized Simple Blinded Study Comparing Two Conversion Ratios From Parenteral to Oral Methadone in Patients With Cancer Pain.
Brief Title: Conversion From Parenteral to Oral Methadone.
Acronym: RATIOMTD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: L'Hospitalet de Llobregat (Other)
Collaborators: Hospital Arnau de Vilanova (Other); Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, JESÚS GONZÁLEZ BARBOTEO, MEDICAL DOCTOR, L'Hospitalet de Llobregat
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RATIOMTD-010810; 2010-024092-39 (EudraCT Number); EC10-133 (Other Grant/Funding Number: Spanish Ministry of Health 2010 Non-Commercial Research Call)
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: Methadone; Pain; Neoplasms; Ratio
MeSH Terms: conditions — Pain; Neoplasms | interventions — Injections; Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parenteral /oral methadone ratio 1:2 (Active Comparator): Far advanced cancer patients with cancer pain hospitalized, and treated with PMTD undergo a preliminary 48 hours observation phase.
  Blinded evaluators assess pain management and treatment toxicity and determine an OPTIMISED DOSE of parenteral METHADONE (pain control without toxicity) for each patient.
  Only patients with a correct control of pain and without significant toxicity throughout this period are eligible for randomization.
  INTERVENTION: Patients randomized to this arm will receive the double of OPTIMISED DOSE of parenteral METHADONE, orally every 24h in 3 administrations during the following 3 days.
  Interventions: Drug: Parenteral /oral methadone ratio 1:2
- Parenteral /oral methadone ratio 1:1.2 (Experimental): Far advanced cancer patients with cancer pain hospitalized, and treated with PMTD undergo a preliminary 48 hours observation phase.
  Blinded evaluators assess pain management and treatment toxicity and determine an OPTIMISED DOSE of parenteral METHADONE (pain control without toxicity) for each patient.
  Only patients with a correct control of pain and without significant toxicity throughout this period are eligible for randomization.
  INTERVENTION: Patients randomized to this arm will receive the following Oral Methadone dose: 20% increase of optimised parenteral methadone dose every 24h in 3 administrations during the following 3 days.
  Interventions: Drug: Parenteral /oral methadone ratio 1:1.2

INTERVENTIONS:
Drug: Parenteral /oral methadone ratio 1:2 — See "arm/group descriptions"
  Other Names: Eptadone (1mg/ml) oral solution
  Arms: Parenteral /oral methadone ratio 1:2
Drug: Parenteral /oral methadone ratio 1:1.2 — See "arm/group descriptions"
  Other Names: Eptadone (1mg/ml) oral solution
  Arms: Parenteral /oral methadone ratio 1:1.2

SUMMARY:
The majority of current studies regarding the use of methadone (MTD) in the treatment of cancer pain are focused in its administration via the oral route (PO). The ratio considered from VO to parenteral route (BP) is 2:1. Academic literature assumes the ratio from BP to VO to be 1:2. In our unit, we use MTD in the context of ROP and not as the last opioid. If face with a situation where there is a good control of pain with MTD BP, usually we move to VO. We have observed that the traditional ratio tend to produce certain toxicity problems. Because of this, we have proposed a new ratio of conversion from PAR MTD to oral MTD, i.e. 1:1.2

DETAILED DESCRIPTION:
OBJECTIVE: To compare the different ratios of conversion from MTD VP to MTD PO. To verify the presence of lower toxicity in the ratio 1:1.2 against 1:2 while still maintaining a good control of pain in patients with advanced cancer that are hospitalized in different palliative care units.

METHODOLOGY: Prospective randomized single blind study in patients with cancer pain treated with parenteral MTD and that would move into MTD oral provided there is good control of pain. The patients will be randomly split into two groups: (Group A = ratio 1:1.2 and Group B=ratio 1:2). Patients will be evaluated during the two days before the switch is applied, the day of the change and during the 3 days post-ROP. The patients who display significant toxicity and/or bad analgesic control within the first 72 hours post-ROP will be considered negative cases. The size of the sample required will include 44 patients distributed in balanced groups in order to obtain a size effect of 45% and a statistical power of 80%. The significance level will be 0.05 for two tails.

STATISTIC ANALYSIS: By means of Chi-squared to compare the proportion of Opioid Rotation (OR) failure in both groups of study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of advanced disease of any type of malignancy;
* >18 years old at the time of inclusion;
* for inclusion in the screening phase, the patient is a candidate to pass parenteral methadone to oral methadone (MTD) following to the physician criteria.
* for inclusion in the assessment phase should follow: presence of cancer pain controlled with no significant toxicity with MTD VP for 48h. Be considered controlled pain and absence of significant toxicity due to MTD, as the definitions given in the general protocol;

  e) signing the informed consent form.

Exclusion Criteria:

1. impairment cognitive status that interferes with the assessment;
2. diagnosis of psychiatric disorders at the time of recruitment that alters the ability to evaluate;
3. presence of side effects due to chemotherapy and / or radiotherapy prior to the change of route of administration, taking into account the following two criteria:

   * For patients on a protocol of successive cycles of chemotherapy (no change in chemotherapy regimen), having presented side effects due to chemotherapy in the 15 days prior to the change of route of administration as clinically and following the recommendations of the 2011 4th ed Oncomecum of the Spanish Society of Medical Oncology and deemed that may interfere with the assessment of the primary endpoint.
   * For patients starting a new protocol of chemotherapy or radiotherapy, have submitted side effects due to such treatment in the 28 days prior to the change of route of administration based on clinical judgment and following the recommendations of the Oncomecum 2011 4th ed. of the Spanish Society of Medical Oncology and deemed that may interfere with the assessment of the primary endpoint.
4. invasive anesthesic techniques have been made during the 3 days before changing to oral parenteral;
5. patients at agony.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of intoxicated patients in each groups | at 3 days after opioid rotation to Oral Methadone

SECONDARY OUTCOMES:
Parenteral/oral MTD final ratio in patients considered as "failure" | One week after the change from pareteral to oral MTD

CONTACTS AND LOCATIONS:
Overall Officials: JESÚS GONZÁLEZ-BARBOTEO, MD, Principal Investigator — INSTITUT CATALÀ D'ONCOLOGIA. HOSPITAL DURAN I REYNALS
Locations (3):
- Spain (3):
  - Institut Català D'Ncologia. Hospital Duran Y Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Background] Gonzalez-Barboteo J, Porta-Sales J, Sanchez D, Tuca A, Gomez-Batiste X. Conversion from parenteral to oral methadone. J Pain Palliat Care Pharmacother. 2008;22(3):200-5. doi: 10.1080/15360280802251199. PMID 19042849